CLINICAL TRIAL: NCT01687400
Title: Genomic Predictors of Decitabine Response in AML/MDS
Brief Title: Genomic Predictors of Decitabine Response in Patients With Acute Myeloid Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201210102
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine (Experimental): Patients receive decitabine IV over 1 hour on days 1-10 of a 28-day cycle. Treatment continues for 2 cycles. Patients then receive decitabine IV over 1 hour on days 1-10, 1-5, or 1-3 (depending on response). Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: decitabine
  Other Names: 5-aza-dCyd, 5AZA, DAC, Dacogen, deoxyazacytidine, dezocitidine

SUMMARY:
This clinical trial studies potential genetic markers which might be used to predict which patients with acute myeloid leukemia or myelodysplastic syndromes respond to decitabine. This study will contribute to the efforts to find effective and less toxic therapies to provide durable remissions in a significant proportion of elderly AML patients.

ELIGIBILITY:
Inclusion Criteria:

All of the following:

* Patient must have non-M3 AML or MDS
* An adverse risk karyotype defined by:

  * Complex karyotype by cytogenetics, or
  * Deletion of all or part of chromosome 5, 7, 12, or 17 defined by FISH or cytogenetics, or
  * Somatic TP53 mutation

All of the following:

1. Patient must have an ECOG performance status ≤ 2.
2. Patient must have >10% disease burden measured by cytomorphology, flow cytometry, or cytogenetics.
3. Patient must have peripheral white blood cell count < 50,000/mcl.
4. Patient must have adequate organ function, defined as:

   1. Total bilirubin < 1.5 x ULN
   2. AST/ALT < 2.5 x ULN
   3. Serum creatinine < 2.0 x ULN
5. Patient must have undergone ≤ 2 cycles of prior hypomethylating agent (decitabine or azacitidine).
6. Patient must be enrolled in HRPO# 201011766 ("Tissue Acquisition for Analysis of Genetic Progression Factors in Hematologic Diseases").
7. Patient must be > 18 years of age.
8. Patient must be able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Patient must not be pregnant or nursing
* Patient must not have acute promyelocytic leukemia or t(15;17) observed by FISH.
* Patient must not have known central nervous system (CNS) leukemia
* Patient must not have a history of positive human immunodeficiency virus (HIV) serology
* Patient must not have a history of positive hepatitis C serology
* Patient must not have undergone prior allogeneic stem cell transplant
* Patient must not have any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, ongoing or active graft-versus-host disease (GVHD), congestive heart failure of New York Heart Association (NYHA) class 3 or 4, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Patient must not have had radiation therapy within 14 days of enrollment
* Patient must not have received any chemotherapy within 21 days of enrollment and any acute treatment-related toxicities must have returned to baseline. Patients may be receiving hydrea at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-02-12 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Welch John, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Welch JS, Petti AA, Miller CA, Fronick CC, O'Laughlin M, Fulton RS, Wilson RK, Baty JD, Duncavage EJ, Tandon B, Lee YS, Wartman LD, Uy GL, Ghobadi A, Tomasson MH, Pusic I, Romee R, Fehniger TA, Stockerl-Goldstein KE, Vij R, Oh ST, Abboud CN, Cashen AF, Schroeder MA, Jacoby MA, Heath SE, Luber K, Janke MR, Hantel A, Khan N, Sukhanova MJ, Knoebel RW, Stock W, Graubert TA, Walter MJ, Westervelt P, Link DC, DiPersio JF, Ley TJ. TP53 and Decitabine in Acute Myeloid Leukemia and Myelodysplastic Syndromes. N Engl J Med. 2016 Nov 24;375(21):2023-2036. doi: 10.1056/NEJMoa1605949. PMID 27959731
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 02/12/2013 and closed to participant enrollment on 06/19/2017.
Period: Overall Study
Arm/Group | Decitabine
Started | 114
Completed | 114
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine
Number analyzed (Participants) | 114
Age, Continuous [Median (Full Range); unit: years] | 73 [31 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 105
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 114

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Patient Specific Mutations With Overall Response Rate
Description: -Best response after 4 treatment cycles as assessed according to International Working Group (IWG) criteria; bone marrow for gene sequencing will be collected at baseline; mutations will be correlated with overall response rate
  --Complete remission (CR), Complete remission with incomplete hematologic recovery (CRi), Marrow complete remission (mCR), Partial remission (PR), Stable disease (SD), Progressive disease (PD)
Time Frame: 4 months (4 treatment cycles)
Population: -Some participants were not evaluable for this outcome measure due to sample collection quality issues and if they had repeat bone marrow biopsies and could be evaluated for responses.
Measure: Count of Participants; unit: Participants
Groups:
- Decitabine (Participants With Response of CR/CRi/mCR/PR); Decitabine (Participants With Response of SD/PD): Patients receive decitabine IV over 1 hour on days 1-10 of a 28-day cycle. Treatment continues for 2 cycles. Patients then receive decitabine IV over 1 hour on days 1-10, 1-5, or 1-3 (depending on response). Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Decitabine (Participants With Response of CR/CRi/mCR/PR) | Decitabine (Participants With Response of SD/PD)
Number analyzed (Participants) | 64 | 22
Participants
  TP53: number analyzed (Participants) | 64 | 17
  TP53 | 26 | 3
  ASXL1: number analyzed (Participants) | 64 | 17
  ASXL1 | 9 | 2
  SRSF2: number analyzed (Participants) | 64 | 17
  SRSF2 | 7 | 5
  IDH2: number analyzed (Participants) | 64 | 17
  IDH2 | 6 | 5
  DNMT3A: number analyzed (Participants) | 64 | 17
  DNMT3A | 8 | 5
  SF3B1: number analyzed (Participants) | 64 | 17
  SF3B1 | 7 | 0
  RUNX1: number analyzed (Participants) | 45 | 15
  RUNX1 | 5 | 3
  TET2: number analyzed (Participants) | 45 | 15
  TET2 | 4 | 3
  IDH1: number analyzed (Participants) | 64 | 17
  IDH1 | 2 | 3
  NPM1: number analyzed (Participants) | 45 | 15
  NPM1 | 4 | 1
  NRAS: number analyzed (Participants) | 45 | 15
  NRAS | 3 | 3
  U2AF1: number analyzed (Participants) | 64 | 17
  U2AF1 | 4 | 1
  MY05B: number analyzed (Participants) | 45 | 15
  MY05B | 3 | 2
  WT1: number analyzed (Participants) | 45 | 15
  WT1 | 5 | 1
Statistical Analysis 1: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #1 is for the genetic mutation TP53; Test type: Other; p = 0.035, Fisher Exact
Statistical Analysis 2: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #2 is for ASXL1 genetic mutation; Test type: Other; p = 0.72, Fisher Exact
Statistical Analysis 3: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #3 is for SRSF2 genetic mutation; Test type: Other; p = 0.28, Fisher Exact
Statistical Analysis 4: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #4 is for IDH2 genetic mutation; Test type: Other; p = 0.14, Fisher Exact
Statistical Analysis 5: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #5 is for DNMT3A genetic mutation; Test type: Other; p = 0.3, Fisher Exact
Statistical Analysis 6: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #6 is for SF3B1 genetic mutation; Test type: Other; p = 0.183, Fisher Exact
Statistical Analysis 7: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #7 is for RUNX1 genetic mutation; Test type: Other; p = 0.42, Fisher Exact
Statistical Analysis 8: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #8 is for TET2 genetic mutation; Test type: Other; p = 0.36, Fisher Exact
Statistical Analysis 9: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #9 is for IDH1 genetic mutation; Test type: Other; p = 0.1, Fisher Exact
Statistical Analysis 10: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #10 is for NPM1 genetic mutation; Test type: Other; p = 1, Fisher Exact
Statistical Analysis 11: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #11 is for NRAS genetic mutation; Test type: Other; p = 0.17, Fisher Exact
Statistical Analysis 12: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); -Statistical analysis #12 is for U2AF1 genetic mutation; Test type: Other; p = 1, Fisher Exact
Statistical Analysis 13: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #13 is for MY05B genetic mutation; Test type: Other; p = 0.6, Fisher Exact
Statistical Analysis 14: Comparison: Decitabine (Participants With Response of CR/CRi/mCR/PR) vs Decitabine (Participants With Response of SD/PD); Statistical analysis #14 is for WT1 genetic mutation; Test type: Other; p = 1, Fisher Exact

2. Secondary Outcome: Compare Outcomes of a 10-day Decitabine Per Cycle Regimen to a 5-day Regimen (Historical Controls)
Description: The overall response rate (CR/CRi/mCR/PR) and complete response rate (CR/CRi/mCR) will be compared with historical controls. Response assessed according to IWG criteria.
Time Frame: 4 months (4 treatment cycles)
Population: -Participants were evaluable for this outcome measure if they completed at least one cycle of treatment and the cycle 1 day 28 bone marrow biopsy to assess response
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Decitabine
Number analyzed (Participants) | 98
percentage of participants
  Overall response rate (CR, CRi/mCR/PR) | 74.42 [65.20 to 83.64]
  Complete response rate (CR, CRi, mCR) | 63.95 [53.81 to 74.10]
Statistical Analysis 1: Comparison: Decitabine; -The historical control of a 5-day regimen (Cashen et al 2010 JCO = NCT00358644) showed 25% (14 out of 55 participants) in overall response rate; Test type: Superiority; p < 0.0001, Chi-squared; 1-sample Chi-square test to compare the overall response rate (ORR) to historical control (with ORR=0.25); Overall Response Rate-for current study = 0.744, 95% CI 2-sided [0.652 to 0.836]
Statistical Analysis 2: Comparison: Decitabine; -The historical control of a 5-day regimen (Cashen et al 2010 JCO = NCT00358644) showed 24% (13 out of 55 participants) in complete response rate; Test type: Superiority; p < 0.0001, Chi-squared; 1-sample Chi-square test to compare the complete response rate to historical control (with CR=0.24); Complete response rate-for current study = 0.640, 95% CI 2-sided [0.538 to 0.741]

3. Secondary Outcome: Rate of Mutation Clearance During Treatment
Description: Samples collected at baseline and after 10, 28 and 56 days of therapy; the rate of mutation clearance was measured as mean VAF change per day of treatment and was estimated using linear mixed model for repeated measurement data .
Time Frame: Up to Day 56
Population: -The first 39 cases with adequate samples were serially evaluated with enhanced exome sequencing. The investigators evaluated 15 additional cases using gene panel sequencing.
Measure: Mean (Standard Deviation); unit: proportion of variant alleles per day
Arm/Group | Decitabine
Number analyzed (Participants) | 54
proportion of variant alleles per day
  TP53: number analyzed (Participants) | 16
  TP53 | -0.781 (0.4423)
  SRSF2: number analyzed (Participants) | 10
  SRSF2 | -0.2214 (0.2705)
  DNMT3A: number analyzed (Participants) | 10
  DNMT3A | -0.2122 (0.2817)
  IDH2: number analyzed (Participants) | 9
  IDH2 | -0.08344 (0.2841)
  RUNX1: number analyzed (Participants) | 8
  RUNX1 | -0.2641 (0.6536)
  TET2: number analyzed (Participants) | 9
  TET2 | -0.07478 (0.3164)
  ASXL1: number analyzed (Participants) | 7
  ASXL1 | -0.3898 (0.3791)
  IDH1: number analyzed (Participants) | 5
  IDH1 | -0.1103 (0.196)
  NRAS: number analyzed (Participants) | 5
  NRAS | 0.04544 (0.2554)
  SF3B1: number analyzed (Participants) | 5
  SF3B1 | -0.719 (0.3481)

4. Secondary Outcome: Peripheral Blood Decitabine Plasma Levels
Description: * To determine whether steady state serum concentrations of decitabine correlated with responses
  * Complete remission (CR), Complete remission with incomplete hematologic recovery (CRi), Partial remission (PR), Stable disease (SD), Progressive disease (PD), Not applicable (NA) - assessed according to International Working Group (IWG) criteria
Time Frame: Day 4
Population: The first 45 participants enrolled with adequate samples were analyzed using GC-MS quantification of serum decitabine levels. Sufficient funds were lacking to complete the analysis of additional participants and all participants with data analyzed are reported.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Decitabine
Number analyzed (Participants) | 45
ng/ml
  CR: number analyzed (Participants) | 3
  CR | 140.5 (53.41)
  CRi: number analyzed (Participants) | 16
  CRi | 117.2 (54.6)
  PR: number analyzed (Participants) | 5
  PR | 67.71 (56.18)
  SD: number analyzed (Participants) | 12
  SD | 145 (73.06)
  PD: number analyzed (Participants) | 3
  PD | 298.5 (213.3)
  NA: number analyzed (Participants) | 6
  NA | 99.64 (58.4)

5. Secondary Outcome: Change in Bone Marrow Methylcytosine
Description: -Change of total bone marrow deoxyribonucleic acid (DNA) methylcytosine from baseline to Day 10
Time Frame: Baseline and Day 10
Measure: Mean (Standard Deviation); unit: proportion of methylcytosine
Groups:
- Decitabine (CR/CRi/mCR); Decitabine (PR/SD/PD): Patients receive decitabine IV over 1 hour on days 1-10 of a 28-day cycle. Treatment continues for 2 cycles. Patients then receive decitabine IV over 1 hour on days 1-10, 1-5, or 1-3 (depending on response). Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Decitabine (CR/CRi/mCR) | Decitabine (PR/SD/PD)
Number analyzed (Participants) | 14 | 11
proportion of methylcytosine
  Day 0 | 0.53 (0) | 0.5374 (0)
  Day 10 | 0.4416 (0.0247) | 0.4639 (0.035)

ADVERSE EVENTS:
Time Frame: -Adverse events were collected from the start of treatment until 30 days following the last day of study treatment (average 5 months) -All deaths were collected from enrollment through study completion date.
Description: Grades 1-5 adverse events will be recorded for the first 50 enrolled participants. Grades 3-5 will be recorded for the remainder of enrolled participants (n=64).
Groups:
- Decitabine (First 50 Enrolled Patients); Decitabine (Remainder of Enrolled Patients n=64): Patients receive decitabine IV over 1 hour on days 1-10 of a 28-day cycle. Treatment continues for 2 cycles. Patients then receive decitabine IV over 1 hour on days 1-10, 1-5, or 1-3 (depending on response). Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Decitabine (First 50 Enrolled Patients) | Decitabine (Remainder of Enrolled Patients n=64)
All-Cause Mortality (participants affected / at risk) | 38/50 | 43/64
Serious Adverse Events (participants affected / at risk) | 42/50 | 47/64
Other Adverse Events (participants affected / at risk) | 50/50 | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (First 50 Enrolled Patients) (N=50) | Decitabine (Remainder of Enrolled Patients n=64) (N=64)
Acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bacteremia - Coagulase negative staphylococcus (Infections and infestations) | 0 | 2
Bacteremia - E. coli (Infections and infestations) | 0 | 2
Bacteremia - ESBL E. coli (Infections and infestations) | 1 | 0
Bacteremia - Enterococcus faecium (Infections and infestations) | 1 | 0
Bacteremia - Klebsiella pneumoniae (Infections and infestations) | 0 | 1
Bacteremia - Micrococcus (Infections and infestations) | 0 | 1
Bacteremia - Staphylococcus capitis (Infections and infestations) | 0 | 1
Bacteremia - Staphylococcus epidermis (Infections and infestations) | 0 | 1
Bacteremia - Staphylococcus infection (Infections and infestations) | 0 | 1
Bacteremia - Streptococcus (Infections and infestations) | 0 | 2
Bacteremia - Streptococcus mitis (Infections and infestations) | 0 | 4
Bacteremia - VRE (Infections and infestations) | 0 | 1
Bacteremia - gram negative (Infections and infestations) | 1 | 0
Bone infection - Osteomyelitis (Infections and infestations) | 1 | 0
C. difficile (Infections and infestations) | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 4 | 2
Cellulitis infection/pneumonia infection (Infections and infestations) | 0 | 1
Central retinal venous occlusion (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 3
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Dental infection (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Diverticulitis infection (Infections and infestations) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Edema (General disorders) | 1 | 0
Endovascular infection (Infections and infestations) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Failure to thrive (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 23 | 30
Fever (General disorders) | 1 | 0
Fusarium fungemia infection (Infections and infestations) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Hematemesis (Gastrointestinal disorders) | 1 | 1
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Iletitis (Infections and infestations) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Infusion related reaction (General disorders) | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Lung infection (Infections and infestations) | 4 | 14
Malaise (General disorders) | 1 | 0
Mucositis - oral (Gastrointestinal disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
NSTEMI (Cardiac disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Parainfluenza infection (Infections and infestations) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Progressive disease/death (General disorders) | 5 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory syncytial virus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
STEMI (Cardiac disorders) | 0 | 2
Sepsis (Infections and infestations) | 3 | 7
Septic arthritis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 3 | 5
Stroke (Nervous system disorders) | 1 | 1
Submandicular sialadenitis infection (Infections and infestations) | 0 | 1
Sweet's syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 3 | 2
Tooth infection (Infections and infestations) | 2 | 0
Upper respiratory infection (Infections and infestations) | 0 | 2
Upper respiratory infection - parainfluenza (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3
White blood cell count decreased (Investigations) | 0 | 1
Bacteremia - Streptococcus mitis/oralis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (First 50 Enrolled Patients) (N=50) | Decitabine (Remainder of Enrolled Patients n=64) (N=64)
Abdominal pain (Gastrointestinal disorders) | 12 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 19 | 5
Acute kidney injury (Renal and urinary disorders) | 7 | 0
Acute renal failure (Renal and urinary disorders) | 0 | 2
Agitation (Psychiatric disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 30 | 2
Alkaline phosphatase increased (Investigations) | 19 | 1
Allergic reaction (Immune system disorders) | 5 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Altered mental status (Psychiatric disorders) | 1 | 0
Anal mucositis (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 14 | 22
Anorexia (Metabolism and nutrition disorders) | 22 | 2
Anxiety (Psychiatric disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 0
Aspartate aminotransferase increased (Investigations) | 26 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 25 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 4
Atrial flutter (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 1
Bacteremia (Gram negative) (Infections and infestations) | 1 | 0
Bacteremia - Escherichia coli/Pseudomonus aeruginosa (Infections and infestations) | 1 | 0
Bacteremia - Myobacterium abscessus (Infections and infestations) | 1 | 0
Bacteremia - Pseudomonas aeruginosa (Infections and infestations) | 1 | 1
Bacteremia - Staphylococcus epidermidis (Infections and infestations) | 2 | 1
Bacteremia - Streptococcus mitis (Infections and infestations) | 0 | 3
Bacteremia - Streptococcus mitis/Coagulase negative staphylococcus (Infections and infestations) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 19 | 0
Blurred vision (Eye disorders) | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone spur (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 21 | 0
Burn (Injury, poisoning and procedural complications) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Burping (Gastrointestinal disorders) | 1 | 0
C. difficile (Infections and infestations) | 2 | 0
Candidal intertrigo (genital) (Infections and infestations) | 1 | 0
Cardiac troponin I increased (Investigations) | 3 | 0
Cardiac troponin T increased (Investigations) | 1 | 0
Catheter related infection (Infections and infestations) | 4 | 6
Chest pain (Cardiac disorders) | 2 | 0
Chills (General disorders) | 31 | 0
Cognitive impairment acute worsening from baseline (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 17 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 25 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 0
Creatinine increased (Investigations) | 8 | 0
Degenerative disc disease (Musculoskeletal and connective tissue disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 15 | 6
Delirium (Psychiatric disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 26 | 0
Diffuse aveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Diverticulitis (Gastrointestinal disorders) | 0 | 2
Diverticulosis (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 15 | 1
Dry eye (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 5 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 | 4
Ear congestion (Ear and labyrinth disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Edema face (General disorders) | 2 | 0
Edema limbs (General disorders) | 31 | 2
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 6 | 3
Encephalopathy (Nervous system disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Esophagitis (Gastrointestinal disorders) | 1 | 0
Facial muscle weakness (Nervous system disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 2
Fatigue (General disorders) | 26 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 13
Fecal incontinence (Gastrointestinal disorders) | 4 | 0
Fever (General disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Floaters (Eye disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 0
Fungal abscess brain (Infections and infestations) | 0 | 1
Fungal infection - spleen and liver (Infections and infestations) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (viral) (Infections and infestations) | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 24 | 6
Gum infection (Infections and infestations) | 1 | 0
HSV infection (Infections and infestations) | 1 | 0
Hallucinations (Psychiatric disorders) | 3 | 0
Hand cramps (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 16 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 2
Hematoma (Skin and subcutaneous tissue disorders) | 5 | 0
Hematuria (Renal and urinary disorders) | 28 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hemorrhage from bronchoscopy (Injury, poisoning and procedural complications) | 0 | 1
Hiatal hernia (Gastrointestinal disorders) | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hip pain following bone marrow biopsy (Injury, poisoning and procedural complications) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hot flashes (Skin and subcutaneous tissue disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 13
Hyperkalemia (Metabolism and nutrition disorders) | 9 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 5 | 1
Hypernatremia (Metabolism and nutrition disorders) | 7 | 1
Hypertension (Vascular disorders) | 2 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 39 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 29 | 1
Hypokalemia (Metabolism and nutrition disorders) | 29 | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 0
Hyponatremia (Metabolism and nutrition disorders) | 37 | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 28 | 13
Hypotension (Vascular disorders) | 14 | 7
Hypothermia (Gastrointestinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 22 | 4
INR increased (Investigations) | 28 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Infection mouth lesion (Infections and infestations) | 1 | 0
Infective myositis (Infections and infestations) | 0 | 1
Infusion related reaction (General disorders) | 9 | 1
Insomnia (Psychiatric disorders) | 9 | 0
Irritability (General disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint infection (Infections and infestations) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 1
Lethargy (Nervous system disorders) | 13 | 0
Localized edema (General disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 17 | 10
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 44 | 45
Lymphocyte count increased (Investigations) | 0 | 1
Malaise (General disorders) | 3 | 0
Mucositis - oral (Gastrointestinal disorders) | 33 | 2
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Nausea (Gastrointestinal disorders) | 28 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 20 | 38
Non-cardiac chest pain (General disorders) | 7 | 0
Oral buccosal infection (Infections and infestations) | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 3 | 1
Oral pain (Gastrointestinal disorders) | 5 | 0
Oral thrush (Infections and infestations) | 13 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pain (General disorders) | 15 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 1
Palpitations (Cardiac disorders) | 2 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 4 | 0
Pericardial tamponade (Cardiac disorders) | 1 | 0
Perineal folliculitis (Infections and infestations) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Photophobia (Eye disorders) | 1 | 0
Platelet count decreased (Investigations) | 27 | 47
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Postoperative hemmorhage (Injury, poisoning and procedural complications) | 3 | 0
Preseptal cellulitis (Infections and infestations) | 0 | 2
Presyncope (Nervous system disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Proteinuria (Renal and urinary disorders) | 22 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 17 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Restless leg syndrome (Nervous system disorders) | 2 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Salivary gland infection (Infections and infestations) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 9 | 1
Septic arthritis (Infections and infestations) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 5 | 0
Sinus pain (Nervous system disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 18 | 0
Sinusitis (Infections and infestations) | 4 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0
Skin infection (Infections and infestations) | 17 | 1
Skin nodules (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 17 | 0
Small bowel obstruction (Gastrointestinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 7 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Stroke (Nervous system disorders) | 1 | 1
Submandibular lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Syncope (Nervous system disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 6 | 2
Tooth infection (Infections and infestations) | 4 | 0
Toothache (Gastrointestinal disorders) | 3 | 1
Tremor (Nervous system disorders) | 2 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 4 | 0
Urinary frequency (Renal and urinary disorders) | 6 | 0
Urinary incontinence (Renal and urinary disorders) | 4 | 0
Urinary retention (Renal and urinary disorders) | 5 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 2 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Ventricular ectopy (Cardiac disorders) | 0 | 1
Vision changes unspecified (Eye disorders) | 1 | 0
Vision loss partial (temporary) (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 19 | 0
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 21 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 | 1
White blood cell decreased (Investigations) | 43 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT01687400/Prot_SAP_000.pdf